CLINICAL TRIAL: NCT05406492
Title: Population Pharmacokinetics of Antibiotics, Sedative and Analgesics, and Antiplatelet Agents During Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: Population PK of Antibiotics, Sedative and Analgesics, and Antiplatelet Drugs During ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Yonsei University (Other)
Responsible Party: Principal Investigator, Jin Wi, Director of Heart Intensive Care Unit, Gachon University Gil Medical Center
Other Study IDs: GDIRB2019-228
Record Dates: First submitted 2022-06-02; First posted 2022-06-06 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Pharmacokinetics; Extracorporeal Membrane Oxygenation
Keywords: Extracorporeal Membrance Oxygenation; Pharmacokinetic medeling; Antiplatelet agents; Sedatives; Antibiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Biospecimen Retention: Samples Without DNA — Residual whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients udergoing ECMO: Population who have been taking antibiotics or antiplatelets or sedatives/analgesics during Extracorporeal Membrane Oxygenation
  Interventions: Other: Residual blood

INTERVENTIONS:
Other: Residual blood — Residual blood samples(1~2 cc) at each sampling time are collected from all subjects while using ECMO for drug concentration assays(LC-MS/MS etc.).

SUMMARY:
The purpose of this study is to optimize the dosage regimen of drugs in patients during during Extracorporeal Membrane Oxygenation (ECMO) by population pharmacokinetic modeling.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are taking levofloxacin, meropenem, vancomycin, cefepime, midalzolam, dexmedetomidine, propofol, clopidogrel, ticagrelor, or prasugrel while underdoing Extracorporeal Membrane Oxygenation

Exclusion Criteria:

* Pregnant women
* Receiving a therapy that can affect blood concentration due to a drug-drug interaction with levofloxacin, meropenem, vancomycin, cefepime, midalzolam, dexmedetomidine, propofol, clopidogrel, ticagrelor, or prasugrel

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are taking levofloxacin, meropenem, vancomycin, cefepime, midalzolam, dexmedetomidine, propofol, clopidogrel, ticagrelor, or prasugrel while underdoing Extracorporeal Membrane Oxygenation
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | Day 0 to day 3 during ECMO, Day 0 to day 3 after removing ECMO
  Volume of distribution
Pharmacokinetic parameters | Day 0 to day 3 during ECMO, Day 0 to day 3 after removing ECMO
  Clearance
Pharmacokinetic parameters | Day 0 to day 3 during ECMO, Day 0 to day 3 after removing ECMO
  Absorption rate (if oral drugs)

CONTACTS AND LOCATIONS:
Locations (1):
- Gacheon University Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shekar K, Fraser JF, Smith MT, Roberts JA. Pharmacokinetic changes in patients receiving extracorporeal membrane oxygenation. J Crit Care. 2012 Dec;27(6):741.e9-18. doi: 10.1016/j.jcrc.2012.02.013. Epub 2012 Apr 18. PMID 22520488
- [Background] Shekar K, Mullany DV, Thomson B, Ziegenfuss M, Platts DG, Fraser JF. Extracorporeal life support devices and strategies for management of acute cardiorespiratory failure in adult patients: a comprehensive review. Crit Care. 2014 May 9;18(3):219. doi: 10.1186/cc13865. PMID 25032748
- [Background] Shekar K, Roberts JA, Welch S, Buscher H, Rudham S, Burrows F, Ghassabian S, Wallis SC, Levkovich B, Pellegrino V, McGuinness S, Parke R, Gilder E, Barnett AG, Walsham J, Mullany DV, Fung YL, Smith MT, Fraser JF. ASAP ECMO: Antibiotic, Sedative and Analgesic Pharmacokinetics during Extracorporeal Membrane Oxygenation: a multi-centre study to optimise drug therapy during ECMO. BMC Anesthesiol. 2012 Nov 28;12:29. doi: 10.1186/1471-2253-12-29. PMID 23190792